CLINICAL TRIAL: NCT00435695
Title: An Open Label, Non-randomized Positron Emission Tomography Study in Healthy Male Subjects to Investigate Brain 5-HT1A Receptor Occupancy, Pharmacokinetics and Safety of Single Oral Doses of GSK163090, Using the Ligand [11C]-WAY100635.
Brief Title: Study Of Safety, Blood Levels, And Brain Receptor Occupancy Of GSK163090 Using PET Imaging In Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTP103265
Record Dates: First submitted 2007-02-13; First posted 2007-02-15 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Subjects; Depressive Disorder and Anxiety Disorders
Keywords: PET scan; healthy males
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — 1-(3-(2-(4-(2-methyl-5-quinolinyl)-1-piperazinyl)ethyl)phenyl)-2-imidazolidinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK163090 (Active Comparator): one infusion only
  Interventions: Drug: GSK163090

INTERVENTIONS:
Drug: GSK163090

SUMMARY:
The purpose of this study is to look at how much of a new drug, GSK163090, binds to proteins in the brain and how much stays in the blood over a range of different doses. This study will use a medical imaging technique called Positron Emission Tomography (PET) which uses an imaging agent called [11C]-WAY100635.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, aged 18-45 years Body weight > 50 kg
* Non-Smoker
* Normal ECG, heart rate and blood pressure

Exclusion Criteria:

* History of any cardiac disease
* History of regular alcohol consumption averaging >14 drinks/week
* Current or recent gastrointestinal disease; History of psychiatric illness including any history of suicidal attempts
* Positive for Hepatitis B and C, and HIV.
* History of drug abuse.
* Exposure to research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden
* Family history of cancer (one or more first-degree relative diagnosed before the age of 55).
* Suffers from claustrophobia
* History or presence of neurological or psychiatric conditions
* Presence of a cardiac pacemaker or other implanted electronic device or metal implants

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Brain receptor occupancy of GSK163090 Plasma concentrations of GSK163090 | throughout the study

SECONDARY OUTCOMES:
Vitals signs ECGs Clinical Laboratory test results | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Toronto, Ontario, Canada